## Examining Engagement Patterns: An Observational Exploration About Tardive Dyskinesia Clinical Trials

An Informed Consent Form For Power Clinical Trial's
Observational Study Involving Patients in Tardive Dyskinesia
Clinical Trials

Date: January 12, 2024

Introduction to the Informed Consent Process: An Overview

This brief summary is designed to offer an overview of our observational clinical study, emphasizing its protocols, potential risks, and benefits for participants. Your consent is a necessity, but your participation is entirely voluntary, granting you the flexibility to withdraw without facing any consequences.

Our study strives to comprehend the factors influencing the decisions of individuals with tardive dyskinesia to join, persist, or discontinue participation in clinical trials. The primary procedures involve the completion of questionnaires and follow-up calls, specifically crafted to minimize potential risks for participants.

While immediate medical benefits may not be evident in this observational study, the amassed data will play a crucial role in identifying strategies to improve clinical trial participation rates, ultimately benefiting those affected by tardive dyskinesia.

The study's outcomes will offer essential insights into the determinants of clinical trial participation rates. Our aim is to enhance recruitment strategies and fortify patient engagement in trials, leading to improved treatment options and outcomes for individuals with tardive dyskinesia. Remember, participation is voluntary, and opting out will not affect your rights.

It is crucial to thoroughly review the consent form and seek clarification on any concerns before making a decision. Engaging in discussions with family, friends, advisors, and healthcare professionals is advisable to ensure an informed choice.

Participation remains completely voluntary, providing the right to withdraw at any time without facing consequences.

Determinants Shaping Involvement in Clinical Trials for Tardive Dyskinesia

While clinical trials play a crucial role in advancing treatments for tardive dyskinesia, questions linger regarding the diverse representation of participants. This investigation delves into the factors influencing patient decisions concerning entry, exit, or re-engagement in clinical trials for tardive dyskinesia. Uncovering these factors is pivotal for enhancing the pertinence and effectiveness of future research endeavors.

To ensure a comprehensive understanding, our focus lies in recruiting a diverse demographic. We seek to unravel how variables like age, race, income, and education shape decisions about participation. The data collected aims to formulate more effective strategies to engage underrepresented groups in upcoming clinical trials.

Participation in this study is entirely voluntary, affording individuals the freedom to withdraw without consequences. The study's procedures, involving questionnaire completion and follow-up calls, pose minimal risks. Prospective participants are strongly urged to thoroughly examine the consent form and seek clarification for any queries.

Ultimately, this trial aims to deepen our understanding of the factors influencing participation in tardive dyskinesia clinical trials. Enhancing participation rates could expedite the development of innovative treatments for this challenging ailment.

Investigating the Participation Behavior of People with Tardive Dyskinesia in Clinical Trials

Our observational clinical study seeks to understand the subtle elements that guide persons with tardive dyskinesia in their clinical trial participation decisions, whether enrollment, withdrawal, or completion. We seek participation in ongoing or completed interventional studies to find potential volunteers, and we use electronic medical data to identify them.

When a participant expresses interest, our staff delivers a detailed permission form outlining the study's aims and participant rights. Regular biweekly questionnaires are used to collect data, which dive into demographics, medical history, and the factors affecting trial participation. In addition, we want to conduct in-depth quarterly phone or video interviews to obtain valuable insights from participants.

The statistical analysis of the collected data aims to reveal the many factors that influence patient involvement in clinical trials. Our findings will be disseminated through conferences and scholarly papers to benefit all parties participating in clinical trials.

These findings will help to shape the design of future clinical trials for people with tardive dyskinesia, as well as enhance recruiting techniques and retention rates.

Participation in this study is fully optional, and subjects have the option to withdraw at any time without penalty. The completion of surveys and follow-up interviews pose few risks, with our easily accessible research staff available to immediately resolve any questions or concerns.

Assessing Risks in Observational Studies of Tardive Dyskinesia

Engaging in observational studies focused on tardive dyskinesia doesn't expose participants to experimental treatments, but it may carry specific risks. These risks could include privacy breaches, emotional distress related to the study's subject matter, and potential adverse outcomes from trial-related procedures.

Prior to committing to participation, it is crucial to thoroughly examine and understand the informed consent form and express any concerns to the research team. The team is committed to providing detailed information about potential risks, the benefits of the study, and the safety measures in place for the protection of participants.

Exploring the Benefits of Participating in Observational Trials for tardive dyskinesia

Involvement in observational clinical trials centered on tardive dyskinesia offers patients an opportunity to play a role in advancing medical knowledge and potentially improving

future treatment options. Despite the absence of experimental therapies, participants can access comprehensive care throughout the study duration.

Prior to making a decision about trial participation, patients are encouraged to meticulously evaluate potential benefits and risks, considering their unique circumstances and goals. Consulting with healthcare providers and the research team becomes crucial in arriving at a well-informed decision.

## Critical Factors Affecting Your Decision to Conclude Participation

Recognizing that your engagement in a clinical trial could conclude without your direct agreement holds considerable importance. Researchers or sponsors might bring the trial to an end for several reasons, such as study suspension, discontinuation of funding, or if it's deemed advantageous for your overall well-being.

Furthermore, your participation might terminate due to deteriorating health, pregnancy, opting out after significant updates, or non-compliance with study guidelines. Deliberating on these elements carefully before committing to clinical trial participation is of utmost significance.

A Comprehensive Look at Different Tardive Dyskinesia Trials

Participation in clinical studies for tardive dyskinesia is fully voluntary, allowing subjects to withdraw without repercussions.

Clinicaltrials.gov, managed by the National Institutes of Health (NIH), is a massive archive of active studies for a complete picture of global <u>research on tardive dyskinesia</u>. Users can tailor their search depending on their region and specific medical issues.

Furthermore, Power's reference page has an up-to-date list of currently ongoing <u>tardive</u> <u>dyskinesia clinical trials</u> that are actively recruiting volunteers.

Exploring the Landscape of Clinical Trial Diversity Online

Several online platforms cater to individuals seeking profound insights into clinical trial diversity. Here are a couple of articles that might capture your interest:

<u>Charrow, Alexandra, Fan Di Xia, Cara Joyce, and Arash Mostaghimi. "Diversity in dermatology clinical trials: a systematic review." *JAMA dermatology* 153, no. 2 (2017): 193-198.</u>

Oh, Sam S., Joshua Galanter, Neeta Thakur, Maria Pino-Yanes, Nicolas E. Barcelo, Marquitta J. White, Danielle M. de Bruin et al. "Diversity in clinical and biomedical research: a promise vet to be fulfilled." *PLoS medicine* 12, no. 12 (2015): e1001918.

These resources provide valuable insights into the challenges associated with clinical trial diversity and potential strategies to foster inclusivity within research studies.

## Safeguarding Privacy in Research Investigations

Our utmost commitment lies in preserving the confidentiality of the data collected for this research endeavor. While complete confidentiality cannot be universally guaranteed, we have instituted robust measures to ensure its protection. It's important to note that legal obligations may, at times, require the disclosure of personal information. Nevertheless, any research publications or presentations will prioritize your anonymity by refraining from revealing your name or any personally identifying information.

Entities such as accrediting bodies, government regulatory authorities (such as the FDA and OHRP), safety monitors, study sponsors, and authorized representatives may access your medical information for purposes related to research, quality assurance, and data analysis.

In exceptional cases, we may request an "Authorization Form" outlining the utilization and sharing of your information for this study. Prior to sharing your information or research samples with Power researchers, other university institutions, or external commercial entities for future research, explicit consent will be sought. Your confidential data will be handled securely and erased as appropriate.

## Consent Acknowledgment: Understanding the Terms

By endorsing this consent agreement, you acknowledge and embrace the following conditions:

 Thoroughly reading and comprehending this informed consent form, with encouragement to explore alternative viewpoints before arriving at a decision.

- Satisfactory resolution of all your inquiries regarding the research project and its methodologies, ensuring you are equipped with the necessary information for study participation.
- Deliberation on potential benefits, drawbacks, and alternatives associated with your involvement in the research.
- Assurance that your voluntary participation in the research study will not impede your legal rights.
- Timely communication of any significant updates that might influence your decision to continue participating in the research study.
- Receipt of this consent form grants you the opportunity to address any lingering inquiries.

| Participant's Signature | | |
|---|---|---|
| Name of Participant | Signature of Participant | Date |
| Confirmation by the Research | her | |
| As the researcher, I have taken the thoroughly, ensuring a compreher reaffirmed that the patient's participation of the comprehensive statement of the comp | nsive understanding of the study. | Furthermore, I have |
| Signature of Researcher Who | o Received Consent | |
| Name of Investigator | Signature of Investigator | <br>Date |